CLINICAL TRIAL: NCT05924945
Title: Impact of Bridge™ Device as a Non-pharmacological Approach to Treat Opioid Withdrawal in Opioid Use Disorder (OUD) Subjects in an Inpatient Treatment Center
Brief Title: Impact of Bridge™ Device to Treat Opioid Withdrawal Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DENE0001
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization table will be kept with the sponsor. Subjects and study site staff (investigators, researchers, care providers) will be blinded to the group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bridge™ active device (Active Comparator): The active Bridge device delivers electrical stimulation to the cranial and occipital nerves.
  Interventions: Device: Bridge™ active device
- Bridge™ sham device (Sham Comparator): The sham device has the same appearance and will require the same placement technique as the Bridge (active) device but will not deliver electrical impulses
  Interventions: Device: Bridge™ sham device

INTERVENTIONS:
Device: Bridge™ active device — Bridge is a percutaneous nerve field stimulation device
  Arms: Bridge™ active device
Device: Bridge™ sham device — The sham device has the same appearance and will require the same placement technique as the Bridge (active) device but will not deliver electrical impulses.
  Arms: Bridge™ sham device

SUMMARY:
The purpose of this prospective study is to investigate the efficacy of the Bridge™ device in reducing the symptoms of opioid withdrawal in a blind comparison to a sham device.

ELIGIBILITY:
Inclusion Criteria:

* Participant able to provide written informed consent
* Participant is 18 to 65-years old
* Participant has confirmed opioid use disorder (OUD) as defined by the Diagnostic and Statistical Manual of Mental Disorders-5
* Participants is entering an OUD treatment program

Exclusion Criteria:

* Participant requires tapering from another substance at entry to treatment
* Participant is pregnant or lactating
* Participant has a history of hemophilia or psoriasis vulgaris
* Participant has a cardiac pacemaker implant device
* Participant has irritated or broken skin at the site of intended device placement
* Participant is currently participating in, or was enrolled in another clinical trial within the last 30 days
* Participant has a history of poor wound healing
* Participant has a severe autoimmune disease or uncontrolled diabetes
* Participant has an open wound/abscess infection/MRSA
* Participant has a history of a chronic pain in the last 90 days
* Participant has a serious medical condition which in the judgment of the principal investigator or his/her designee would make study participation unsafe, or would make intervention compliance difficult
* Participant has a psychiatric illness (bipolar disorder, schizophrenia, or other psychotic disorder, active suicidal ideation with a plan within the last month or suicide attempt)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Caron Treatment Centers, Wernersville, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bridge™ Active Device | Bridge™ Sham Device
Started | 6 | 7
Completed | 3 | 3
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bridge™ Active Device | Bridge™ Sham Device | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 5 | 10
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Assess Change in Clinical Opiate Withdrawal Scale (COWS) Score
Description: The Clinical Opiate Withdrawal Scale (COWS) is an 11-item scale designed to be administered by a clinician. This tool can be used in both inpatient and outpatient settings to reproducibly rate common signs and symptoms of opiate withdrawal and monitor these symptoms over time. The summed score for the complete scale can be used to help clinicians determine the stage or severity of opiate withdrawal and assess the level of physical dependence on opioids. Score Range: The COWS score can range from 0 to 48.
  Interpretation:
  0-4: No withdrawal 5-12: Mild withdrawal 13-24: Moderate withdrawal 25-36: Moderately severe withdrawal 37-48: Severe withdrawal High scores mean more severe withdrawal.
Time Frame: prior to device placement (0 min), 30 min, 60 min, 120 min, 2nd day, 3rd day, 4th day and 5th day of continuous device use
Population: The study was terminated prematurely due to sponsor decision with no clinical rationale for the termination. This was a prospective study investigating the test device. Of 13 subjects using the device, only 6 completed the study. The sample size is well below the threshold needed to perform reliable statistical comparisons. We reported all demographic data and outcome measure data from the limited sample. Further data reporting would be statistically inappropriate due to the sample size.
Measure: Number; unit: score on a scale
Arm/Group | Bridge™ Active Device | Bridge™ Sham Device
Number analyzed (Participants) | 3 | 3
score on a scale
  Subject 1 COWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 COWS score pre-device placement, 0 min device use (raw data) |  | 18
  Subject 1 COWS score device use 30 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 COWS score device use 30 min (raw data) |  | 5
  Subject 1 COWS score device use 60 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 COWS score device use 60 min (raw data) |  | 3
  Subject 1 COWS score device use 120 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 COWS score device use 120 min (raw data) |  | 6
  Subject 1 COWS score device use 2 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 COWS score device use 2 days (raw data) |  | 10
  Subject 1 COWS score device use 3 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 COWS score device use 3 days (raw data) |  | 8
  Subject 1 COWS score device use 4 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 COWS score device use 4 days (raw data) |  | 0
  Subject 1 COWS score device use 5 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 COWS score device use 5 days (raw data) |  | 7
  Subject 2 COWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 COWS score pre-device placement, 0 min device use (raw data) |  | 15
  Subject 2 COWS score device use 30 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 COWS score device use 30 min (raw data) |  | 7
  Subject 2 COWS score device use 60 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 COWS score device use 60 min (raw data) |  | 3
  Subject 2 COWS score device use 120 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 COWS score device use 120 min (raw data) |  | 5
  Subject 2 COWS score device use 2 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 COWS score device use 2 days (raw data) |  | 9
  Subject 2 COWS score device use 3 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 COWS score device use 3 days (raw data) |  | 13
  Subject 2 COWS score device use 4 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 COWS score device use 4 days (raw data) |  | 15
  Subject 2 COWS score device use 5 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 COWS score device use 5 days (raw data) |  | 13
  Subject 3 COWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 COWS score pre-device placement, 0 min device use (raw data) |  | 17
  Subject 3 COWS score device use 30 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 COWS score device use 30 min (raw data) |  | 14
  Subject 3 COWS score device use 60 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 COWS score device use 60 min (raw data) |  | 10
  Subject 3 COWS score device use 120 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 COWS score device use 120 min (raw data) |  | 9
  Subject 3 COWS score device use 2 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 COWS score device use 2 days (raw data) |  | 16
  Subject 3 COWS score device use 3 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 COWS score device use 3 days (raw data) |  | 3
  Subject 3 COWS score device use 4 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 COWS score device use 4 days (raw data) |  | 3
  Subject 3 COWS score device use 5 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 COWS score device use 5 days (raw data) |  | 5
  Subject 4 COWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 COWS score pre-device placement, 0 min device use (raw data) | 16 |
  Subject 4 COWS score device use 30 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 COWS score device use 30 min (raw data) | 8 |
  Subject 4 COWS score device use 60 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 COWS score device use 60 min (raw data) | 6 |
  Subject 4 COWS score device use 120 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 COWS score device use 120 min (raw data) | 5 |
  Subject 4 COWS score device use 2 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 COWS score device use 2 days (raw data) | 4 |
  Subject 4 COWS score device use 3 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 COWS score device use 3 days (raw data) | 6 |
  Subject 4 COWS score device use 4 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 COWS score device use 4 days (raw data) | 5 |
  Subject 4 COWS score device use 5 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 COWS score device use 5 days (raw data) | 3 |
  Subject 5 COWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 COWS score pre-device placement, 0 min device use (raw data) | 20 |
  Subject 5 COWS score device use 30 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 COWS score device use 30 min (raw data) | 7 |
  Subject 5 COWS score device use 60 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 COWS score device use 60 min (raw data) | 7 |
  Subject 5 COWS score device use 120 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 COWS score device use 120 min (raw data) | 2 |
  Subject 5 COWS score device use 2 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 COWS score device use 2 days (raw data) | 4 |
  Subject 5 COWS score device use 3 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 COWS score device use 3 days (raw data) | 2 |
  Subject 5 COWS score device use 4 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 COWS score device use 4 days (raw data) | 1 |
  Subject 5 COWS score device use 5 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 COWS score device use 5 days (raw data) | 0 |
  Subject 6 COWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 COWS score pre-device placement, 0 min device use (raw data) | 16 |
  Subject 6 COWS score device use 30 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 COWS score device use 30 min (raw data) | 11 |
  Subject 6 COWS score device use 60 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 COWS score device use 60 min (raw data) | 10 |
  Subject 6 COWS score device use 120 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 COWS score device use 120 min (raw data) | 8 |
  Subject 6 COWS score device use 2 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 COWS score device use 2 days (raw data) | 8 |
  Subject 6 COWS score device use 3 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 COWS score device use 3 days (raw data) | 8 |
  Subject 6 COWS score device use 4 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 COWS score device use 4 days (raw data) | 9 |
  Subject 6 COWS score device use 5 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 COWS score device use 5 days (raw data) | 4 |

2. Secondary Outcome: Assess Change in Subjective Opiate Withdrawal Scale (SOWS) Score
Description: The Subjective Opiate Withdrawal Scale (SOWS) consist of 16 symptoms rated in intensity by patients on a 5-point scale of intensity as follows: 0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely. The total score is a sum of item ratings, and ranges from 0 to 64.
  High scores mean worse symptom intensity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: score on a scale
Arm/Group | Bridge™ Active Device | Bridge™ Sham Device
Number analyzed (Participants) | 3 | 3
score on a scale
  Subject 1 SOWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 SOWS score pre-device placement, 0 min device use (raw data) |  | 40
  Subject 1 SOWS score device use 30 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 SOWS score device use 30 min (raw data) |  | 42
  Subject 1 SOWS score device use 60 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 SOWS score device use 60 min (raw data) |  | NA — score at this time point not obtained
  Subject 1 SOWS score device use 120 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 SOWS score device use 120 min (raw data) |  | 24
  Subject 1 SOWS score device use 2 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 SOWS score device use 2 days (raw data) |  | 38
  Subject 1 SOWS score device use 3 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 SOWS score device use 3 days (raw data) |  | 28
  Subject 1 SOWS score device use 4 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 SOWS score device use 4 days (raw data) |  | 19
  Subject 1 SOWS score device use 5 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 1 SOWS score device use 5 days (raw data) |  | 28
  Subject 2 SOWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 SOWS score pre-device placement, 0 min device use (raw data) |  | 23
  Subject 2 SOWS score device use 30 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 SOWS score device use 30 min (raw data) |  | 10
  Subject 2 SOWS score device use 60 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 SOWS score device use 60 min (raw data) |  | 10
  Subject 2 SOWS score device use 120 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 SOWS score device use 120 min (raw data) |  | 10
  Subject 2 SOWS score device use 2 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 SOWS score device use 2 days (raw data) |  | 16
  Subject 2 SOWS score device use 3 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 SOWS score device use 3 days (raw data) |  | 19
  Subject 2 SOWS score device use 4 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 SOWS score device use 4 days (raw data) |  | 32
  Subject 2 SOWS score device use 5 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 2 SOWS score device use 5 days (raw data) |  | 34
  Subject 3 SOWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 SOWS score pre-device placement, 0 min device use (raw data) |  | 46
  Subject 3 SOWS score device use 30 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 SOWS score device use 30 min (raw data) |  | 49
  Subject 3 SOWS score device use 60 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 SOWS score device use 60 min (raw data) |  | 35
  Subject 3 SOWS score device use 120 min (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 SOWS score device use 120 min (raw data) |  | 37
  Subject 3 SOWS score device use 2 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 SOWS score device use 2 days (raw data) |  | 43
  Subject 3 SOWS score device use 3 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 SOWS score device use 3 days (raw data) |  | 18
  Subject 3 SOWS score device use 4 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 SOWS score device use 4 days (raw data) |  | 9
  Subject 3 SOWS score device use 5 days (raw data): number analyzed (Participants) | 0 | 1
  Subject 3 SOWS score device use 5 days (raw data) |  | 9
  Subject 4 SOWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 SOWS score pre-device placement, 0 min device use (raw data) | 32 |
  Subject 4 SOWS score device use 30 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 SOWS score device use 30 min (raw data) | 12 |
  Subject 4 SOWS score device use 60 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 SOWS score device use 60 min (raw data) | 10 |
  Subject 4 SOWS score device use 120 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 SOWS score device use 120 min (raw data) | 9 |
  Subject 4 SOWS score device use 2 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 SOWS score device use 2 days (raw data) | 11 |
  Subject 4 SOWS score device use 3 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 SOWS score device use 3 days (raw data) | 11 |
  Subject 4 SOWS score device use 4 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 SOWS score device use 4 days (raw data) | 6 |
  Subject 4 SOWS score device use 5 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 4 SOWS score device use 5 days (raw data) | 5 |
  Subject 5 SOWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 SOWS score pre-device placement, 0 min device use (raw data) | 47 |
  Subject 5 SOWS score device use 30 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 SOWS score device use 30 min (raw data) | 26 |
  Subject 5 SOWS score device use 60 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 SOWS score device use 60 min (raw data) | 22 |
  Subject 5 SOWS score device use 120 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 SOWS score device use 120 min (raw data) | 14 |
  Subject 5 SOWS score device use 2 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 SOWS score device use 2 days (raw data) | 12 |
  Subject 5 SOWS score device use 3 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 SOWS score device use 3 days (raw data) | 10 |
  Subject 5 SOWS score device use 4 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 SOWS score device use 4 days (raw data) | 4 |
  Subject 5 SOWS score device use 5 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 5 SOWS score device use 5 days (raw data) | 4 |
  Subject 6 SOWS score pre-device placement, 0 min device use (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 SOWS score pre-device placement, 0 min device use (raw data) | 36 |
  Subject 6 SOWS score device use 30 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 SOWS score device use 30 min (raw data) | 25 |
  Subject 6 SOWS score device use 60 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 SOWS score device use 60 min (raw data) | 24 |
  Subject 6 SOWS score device use 120 min (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 SOWS score device use 120 min (raw data) | 19 |
  Subject 6 SOWS score device use 2 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 SOWS score device use 2 days (raw data) | 17 |
  Subject 6 SOWS score device use 3 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 SOWS score device use 3 days (raw data) | 11 |
  Subject 6 SOWS score device use 4 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 SOWS score device use 4 days (raw data) | 8 |
  Subject 6 SOWS score device use 5 days (raw data): number analyzed (Participants) | 1 | 0
  Subject 6 SOWS score device use 5 days (raw data) | 6 |

ADVERSE EVENTS:
Time Frame: Through end of study participation (approximately 3 weeks)
Arm/Group | Bridge™ Active Device | Bridge™ Sham Device
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bridge™ Active Device (N=3) | Bridge™ Sham Device (N=3)
Pain (Nervous system disorders) | 0 (0) | 1 (1) — Pain or discomfort at the site of device application

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to sponsor decision with no clinical rationale for termination. This prospective study investigated a test device deemed "end-of-life" by the manufacturer. Only 13 subjects used devices of 48 anticipated; 6 subjects completed the study (3 with active device, 3 with shame device).

We reported all demographic data and outcome measure data from the limited sample size. Further data reporting would be statistically inappropriate due to the sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Rev B (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT05924945/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Rev A (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT05924945/Prot_SAP_002.pdf